CLINICAL TRIAL: NCT02173210
Title: Precision Medicine In Segregating Endotypes in Preterm Birth
Brief Title: Precision Medicine for Preterm Birth
Acronym: PRoMISE
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 820143
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Premature Birth
Keywords: Premature birth; Premature delivery; Metabolomics; Microbiota; Genetics; 17 hydroxyprogesterone caproate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prior preterm birth: Pregnant women with a prior preterm birth, eligible to receive 17 hydroxyprogesterone caproate (17OHPC)

SUMMARY:
This project is examining genetic and metabolic markers for the use of 17 hydroxyprogesterone caproate (17OHPC) in pregnant women with a history of preterm birth (PTB). 17OHPC has been associated with a 30-35% reduction in repeat PTB in women carrying a singleton gestation. However, it is not well known why it works for some women but not for others. There are limited available interventions for the prevention of recurrent PTB. This study will enroll 150 women at risk for PTB and eligible to receive 17OHPC, and expect that 80% will use 17OHPC and 20% will decline use. We will obtain blood samples and samples of cervical cells and cervical vaginal fluid. The objective of the study is to identify genetic, microbial and molecular markers that help to identify which women at risk for recurrent preterm birth will respond to 17OHPC and which women will not. The ultimate goal is to develop a personalized screening test based on these markers.

DETAILED DESCRIPTION:
Women with a prior preterm birth will be recruited between 16 and 22 weeks gestation. At this initial time point, samples of cervical epithelial cells and cervicovaginal fluid will be collected. Approximately 8 weeks later, those samples will be collected a second time, along with a blood sample. Outcome data will be collected after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women with a prior spontaneous preterm birth of a singleton pregnancy (delivered at 16-36 6/7 weeks gestation)
* Singleton in the current pregnancy
* Eligible to use 17 hydroxyprogesterone caproate (17OHPC) in this pregnancy for clinical indications
* 16-22 weeks gestation at the time of visit 1 assessments

Exclusion Criteria:

* Major fetal anomaly
* Allergy to 17OHPC

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with a singleton gestation who have had a prior spontaneous preterm birth.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Preterm Birth | At time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Michal Elovitz, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania